CLINICAL TRIAL: NCT01591629
Title: Assessment of Cannabinoid-opiate Interactions in Humans With a Cannabis Use Disorder and Healthy Subjects
Brief Title: The Effects of ∆-9-THC and Naloxone in Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Associate Professor, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1108008940
Record Dates: First submitted 2012-04-25; First posted 2012-05-04 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: Cannabis; Marijuana; Naloxone; THC; Psychotic Disorders
MeSH Terms: conditions — Marijuana Abuse; Psychotic Disorders | interventions — Naloxone; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo and Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Active Naloxone and Placebo (Experimental)
  Interventions: Drug: Naloxone; Drug: Placebo
- Placebo and Active Delta-9-THC (Placebo Comparator)
  Interventions: Drug: Delta-9-THC; Drug: Placebo
- Active Naloxone and Active Delta-9-THC (Experimental)
  Interventions: Drug: Naloxone; Drug: Delta-9-THC

INTERVENTIONS:
Drug: Naloxone — Active Naloxone 18 mcg/kg intravenously over 60 minutes, 2mg IV push, 1mg IV push
  Arms: Active Naloxone and Active Delta-9-THC; Active Naloxone and Placebo
Drug: Delta-9-THC — Active Delta-9-THC (0.025mg/Kg) given intravenously over 20 minutes.
  Arms: Active Naloxone and Active Delta-9-THC; Placebo and Active Delta-9-THC
Drug: Placebo — Placebo
  Arms: Active Naloxone and Placebo; Placebo and Active Delta-9-THC; Placebo and Placebo

SUMMARY:
The purpose of this project is to examine the effects of mu-opiate antagonism on the rewarding and reinforcing effects of delta-9-tetrahydrocannabinol (THC), the main psychoactive ingredient of cannabis.

ELIGIBILITY:
Inclusion Criteria:

* At least one exposure to Cannabis

Exclusion Criteria:

* Cannabis Naive

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-11-04 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2012-06-01 (Actual)

PRIMARY OUTCOMES:
Behavioral Measures | 4 test days
  Subjective effects and perceptual alterations will be assessed using the Positive and Negative Symptom Subscale (PANNS).

SECONDARY OUTCOMES:
Visual analog scales | 4 test days
  Will assess subjective effects, perceptual alterations, and cognitive effects.
Clinician Administered Dissociative States Scales (CADSS) | 4 test days
  Will measure subjective effects, perceptual alterations, and cognitive effects.
Psychotomimetic States Inventory (PSI) | 4 test days
  Will assess subjective effects, perceptual alterations, and cognitive effects.
Marijuana Withdrawal Scale | 4 test days
  Will assess subjective effects, perceptual alterations, and cognitive effects.
Clinical Opiate Withdrawal Scale | 4 test days
  Will assess subjective effects, perceptual alterations, and cognitive effects.
Marijuana Craving Scale | 4 test days
  Will assess subjective effects, perceptual alterations, and cognitive effects.
Neuro cognitive battery | 4 test days
  Will assess cognitive effects.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States